CLINICAL TRIAL: NCT06900582
Title: Comparing SENTInel Node Mapping to Comprehensive Lymphadenectomy in P53-Mutated EndoMETRial Cancer: a Prospective, Open-label, Controlled, Randomized, Non-inferiority, De-escalation Trial
Brief Title: SENTInel Node Mapping Versus Comprehensive Lymphadenectomy in P53-Mutated Endometrial Cancer: a Non-Inferiority Randomized Trial
Acronym: SENTIMETREP53
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9423
Record Dates: First submitted 2025-03-10; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Lymphadenectomy; Endometrial Cancer; Gene, P53; Sentinel Lymph Node Biopsy (SLNB)
Keywords: Endometrial cancer; Sentinel lymph node biopsy; Lymphadenectomy; p53 mutation
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sentinel Lymph Node Mapping (Experimental): Patients in this arm will undergo sentinel lymph node (SLN) mapping, followed by total hysterectomy, bilateral salpingo-oophorectomy, and, for serous, carcinosarcoma and undifferentiated type EC, infracolic omentectomy. The determination to perform para-aortic lymphadenectomy on SLN+ patients is left to the clinical team. Adjuvant treatment will depend of the status.
  Interventions: Procedure: Sentinel Lymph Node Mapping
- Complete lymphadenectomy (Active Comparator): Patients in this arm will undergo comprehensive pelvic and para-aortic lymphadenectomy that extends up to the left renal vein, followed by total hysterectomy and bilateral salpingo-oophorectomy, with omentectomy for serous, carcinosarcoma and undifferentiated type EC. Adjuvant treatment will depend of the status.
  Interventions: Procedure: Comprehensive pelvic and para-aortic lymphadenectomy

INTERVENTIONS:
Procedure: Sentinel Lymph Node Mapping — The SLN mapping protocol will follow the EU guidelines and the consensus in competency assessment tool. Prior to SLN mapping, a full inspection of the pelvic areas with white light is performed to exclude the presence of extrauterine disease. The next surgical steps will be 1- identification of external iliac vessels, 2- identification of internal iliac artery, 3- dissection of the ureter, 4- development of paravesical space and 5- identification of obliterated umbilical ligament. The dissection technique must avoid disrupting lymphatic channels and isolate nodal tissue from the local anatomy. Indocyanine green (1.25mg/mL) will be injected in the cervix at the 3 and 9 o'clock positions, with 1mL superficial and 1mL deep, for a total of 4mL. All mapped SLNs must be completely excised, and any visually suspicious nodes should also be removed, regardless of the mapping results. If the SLN mapping appears to be unfeasible, a side-specific pelvic lymphadenectomy will be performed.
  Arms: Sentinel Lymph Node Mapping
Procedure: Comprehensive pelvic and para-aortic lymphadenectomy — The resection of at least one lymph node in each of the 12 retroperitoneal regions is necessary:
  A: upper para-aortic region B: lower para-aortic region C: interaorto-caval region D: paracaval region E: right and left iliaca communis region F: right and left iliaca externa region G: right and left fossa obturatoria region: defined by external and internal arteria iliaca, pelvic sidewall H: right and left iliaca interna region: lymph nodes adjacent to or medial of the internal iliacal artery
  Arms: Complete lymphadenectomy

SUMMARY:
This study evaluates surgical strategies for treating patients with FIGO 2023 stage I and II high-risk endometrial cancer (EC) exhibiting p53 mutations. The trial aims to assess whether a less invasive sentinel lymph node (SLN) mapping approach provides non-inferior oncological outcomes compared to the current standard of systematic pelvic and para-aortic lymphadenectomy (PL+PALND). By minimizing surgical morbidity, this study seeks to determine if SLN mapping can safely replace comprehensive lymphadenectomy without compromising disease-free survival (DFS). Eligible patients will be randomized to undergo either sentinel lymph node mapping or complete lymphadenectomy, followed by standard hysterectomy and bilateral salpingo-oophorectomy. The primary outcome is DFS at 36 months, with secondary outcomes including overall survival, disease-specific survival, perioperative complications, and quality of life.

DETAILED DESCRIPTION:
The necessity of extensive lymph node dissection in endometrial cancer remains a subject of debate. Although systematic pelvic and para-aortic lymphadenectomy (PL+PALND) improves disease staging and influences adjuvant therapy, its impact on survival in high-risk endometrial cancer (EC) is still controversial. Recent evidence suggests that SLN mapping may provide comparable staging accuracy while reducing surgical complications. However, the oncological safety of replacing PL+PALND with SLN mapping in high-risk EC patients, particularly those with p53 mutations, remains uncertain.

This study is designed as a prospective, multicenter, randomized controlled trial to evaluate the non-inferiority of SLN mapping versus PL+PALND in patients with high-risk EC characterized by p53 mutations. Patients will be stratified based on tumor histology and imaging findings before undergoing surgery. The trial will enroll 374 patients across 22 participating centers.

Key issues addressed include:

* Oncological Safety: Assessing whether SLN mapping provides equivalent DFS compared to PL+PALND.
* Survival Outcomes: Evaluating overall survival (OS) and disease-specific survival (DSS) at 36 months.
* Surgical Morbidity: Comparing perioperative and postoperative complications
* Quality of Life: Determining patient-reported outcomes related to surgical recovery and long-term functional status.

This study integrates modern molecular classifications, recognizing p53 mutations as a significant prognostic marker. If SLN mapping is proven non-inferior, it could lead to a paradigm shift, reducing the extent of surgical intervention for high-risk EC patients while maintaining oncological safety.

ELIGIBILITY:
Inclusion Criteria:

1 . ≥ 18 years old 2. High-risk endometrial cancer, as defined by the ESGO-ESTRO 20211 histological and molecular classification, with p53 mutation confirmed on endometrial biopsy or curettage in the two months before the surgery 3. Magnetic Resonance Imaging (MRI) confirmed FIGO 2023 stage I and II endometrial cancer, i.e., confined to the uterine corpus, ovary and the cervical stroma.

4. Participant with a scheduled surgical intervention (total hysterectomy and bilateral salpingo-oophorectomy, with omentectomy in the case of serous, carcinosarcoma and undifferenciated type EC) 5. Eligible for comprehensive lymphadenectomy by laparoscopy 6. Participant with a negative Positron Emission Tomography scan (PET-CT scan) for lymph node involvement in the two months before the intervention 7. ECOG (Eastern Cooperative Oncology Group) performance status of 0-1 8. Participant able to provide written informed consent

Exclusion Criteria:

1. Recurrent EC
2. Previous chemo-, radio, or endocrine therapy for EC
3. Any contra-indication to lymphadenectomy and/or chemotherapy
4. Any contraindication to laparoscopy
5. Any criteria, based on the investigator's judgment, that would contraindicate the surgical procedure (e.g., but not limited to, anesthetic risk, bleeding, significant comorbidities)
6. Any known disorder or circumstances making participation in trial and follow-up questionable
7. Patients with other malignancies for whom the disease(s) and/or associated treatment(s) might have an impact on the patient's cancer prognosis
8. Known HIV-infection or AIDS
9. Simultaneous participation in another interventional clinical trial
10. Within the exclusion period following participation in another interventional clinical trial
11. Patients with difficulties in reading or understanding French, or an inability to understand the delivered information
12. Patients in emergency medical situations
13. Patient under guardianship or limited guardianship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2031-10 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
Disease-free-survival (DFS) | 36 months
  Time from randomization to first recurrence or death from any cause, censored at last follow-up

SECONDARY OUTCOMES:
Overall survival (OS) | 36 months
  Time from randomization to death due to endometrial cancer, censored for other deaths/last follow-up.
Disease-specific survival (DSS) | 36 Months
  Time from randomization to death due to endometrial cancer,
Perioperative complications rate and postoperative complications rate | At 30- and 90-days
  The classification of Clavien-Dindo will be used.
Return to intended oncologic treatment (RIOT) | From the date of surgery (Day 0) until the first day of adjuvant treatment, assessed up to 90 days.
  Time in days between the date of surgery and the first day of adjuvant treatment.
Quality of life - EORTC QLQ-C30 questionnaire score | At baseline, 1, 6 and 12 months
  EORTC QLQ-C30 questionnaire is a 30 item instrument meant to assess some of the different aspects that define the quality of life of cancer patients
Quality of life - EORTC QLQ-EN24 questionnaire score | At baseline, 1, 6 and 12 months
  EORTC QLQ-EN24 questionnaire is designed to assess disease and treatment specific aspects of the quality of life of patients with endometrial cancer
Accuracy of PET-CT scan in the detection of metastatic lymph nodes | From Day -60 to Day -1 before surgery (Day 0)
  Determination of the sensitivity, specificity, positive and negative predictive value
Assessment of the rate of unsuccessful SLN mapping, requiring conversion to pelvic lymphadenectomy | At surgery time
  Rate of unsuccessful SLN mapping, requiring conversion to pelvic lymphadenectomy